CLINICAL TRIAL: NCT05280405
Title: Impact of Early Proactive Therapeutic Drug Monitoring on the Durability and Efficacy of Infliximab Therapy in Pediatric Inflammatory Bowel Disease: a Multicenter Open-label Randomized-control Trial
Brief Title: Early Proactive Therapeutic Drug Monitoring of Infliximab in Children: EPIC Study
Acronym: EPIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-003220-32
Record Dates: First submitted 2022-02-22; First posted 2022-03-15 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Infliximab; Proactive drug monitoring
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-Proactive Therapeutic Drug Monitoring (E-pTDM) (Experimental): Infliximab (IFX) at 5mg/kg, IV at week 0, 2 and 6. From week 6, the infusion interval will be adjusted based on pre-infusion IFX concentrations to target a trough level grater or equal to (>=) 5 mcg/ml (> 10 μg/ml in patients with perianal disease). For IFX concentrations below target, the infusion interval will be shortened (minimum interval 2 weeks). IFX dose increase will be performed as a second step.
  Interventions: Drug: Infliximab
- Standard dosing (Active Comparator): Infliximab (IFX) at 5mg/kg, IV at week 0, 2 and 6 followed by 5mg/kg infusions every 8 weeks.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab

SUMMARY:
The purpose of the study is to assess whether a proactive therapeutic drug monitoring strategy, introduced early during treatment, improves Infliximab (IFX) durability, efficacy and safety in children and young adults with inflammatory bowel disease. Patients with an indication to receive IFX, based on current clinical practice recommendations, will receive the drug either based on IFX concentrations determined before every IFX infusion, starting from the third infusion, or at standard dosing. Approximately 90 patients will be included in this research study. Patients enrolled will be in the study for approximately 12 months.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) are relapsing disorders with progressive bowel damage leading to long-term disability.

Infliximab (IFX), is a highly effective and commonly used biologic in IBD. However, up to 40% of patients do not respond to treatment or lose response over time. Low-serum IFX concentrations and the development of antibodies to IFX (ATI) are two major factors affecting IFX efficacy, durability and safety. Standard IFX dose is administered as an IV (in the vein) infusion at 5 mg/kg in a 0, 2, and 6 weeks induction regimen followed by a maintenance regimen with infusions every 8 weeks. This standard dosing is extrapolated from adult studies. IFX has a highly variable pharmacokinetic and pharmacodynamics that is dependent on body weight, disease extent, levels of inflammation and the presence of ATI. In children and young adults with IBD all these factors often result in low-serum IFX concentrations.

Proactive therapeutic drug monitoring, consists in the measurement of drug concentrations on patient's blood, in order to adjust the following administrations (dosing or interval) and maintain a desired concentration of the medication in the body.

This study seeks to determine whether a proactive therapeutic drug monitoring strategy can improve IFX durability, efficacy and safety in children and young adults with IBD. The study will involve approximately 90 patients, aged 6 to 17 years, with IBD. All the patients enrolled in the study will receive IFX at 5mg/kg at week 0, 2 and 6. At week 6 patients will be randomly assigned to receive IFX treatment either based on IFX concentrations determined before every IFX infusion (intervention group) or at standard dosing (control group). Patients will participate in the study for 54 weeks (approximately 12 months) or until IFX discontinuation. During the study, patients will visit the study center at the time of every IFX infusion or in case of disease flares.

ELIGIBILITY:
Inclusion Criteria:

1. Anti-TNF naïve children and adolescents, 6-17 years, with a diagnosis of IBD confirmed by a prior endoscopic biopsy that is consistent with the diagnosis
2. Indication to start anti-TNF therapy in accordance with current pediatric guidelines for the treatment of pediatric IBD
3. Active inflammation supported by CRP > 5mg/L and /or FC > 150 μg/g before the 1st IFX dose

Exclusion Criteria:

1. Consent withdrawal,
2. Stenosing or penetrating disease requiring surgery, abdominal abscess, symptomatic stricture,
3. Abdominal surgery within the previous 6 months,
4. Acute severe ulcerative colitis attack defined by a PUCAI score Ñ 65,
5. Infective contraindication to IFX treatment including positive tuberculin skin test or Quantiferon-TB test, recent opportunistic infection, infection with hepatitis B (HBV), C (HCV), human immunodeficiency virus (HIV),
6. Previous exposure to anti-TNF;
7. Exposure to concomitant prohibited medications including other biologics (including but not limited to ustekinumab, vedolizumab, abatacept, anakinra..), thalidomide, investigational drugs
8. Pregnancy or lactation

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of IFX discontinuation or need for treatment intensification due to non-response or LOR during the first year of treatment. | 54 weeks
  Composite outcome. Treatment intensification is defined as adjunction of rescue therapies, including corticosteroids systemic or topical, azathioprine (AZA), methotrexate (MTX), 5-aminosalicylate (5-ASA) systemic or topical, or rescue IFX escalation or surgery; treatment response is defined as a decrease in Pediatric Crohn's Disease Activity Index (PCDAI) by 12.5 point or in Pediatric Ulcerative Colitis Activity Index (PUCAI) by 10 points with decrease in C reactive protein (CRP) by 50% after induction, evaluated between 12-14 weeks; loss of response (LOR) is defined as PCDAI >= 10 or PUCAI > 10 with CRP > 0.5mg/dl and/or fecal calprotectin (FC) >250 microg/g in a patient who previously responded to induction treatment.

SECONDARY OUTCOMES:
Cumulative probability of IFX discontinuation | 54 weeks
  Time to IFX discontinuation
Cumulative probability of Loss of Response | 54 weeks
  Time to Loss of Response (LOR), with LOR defined as PCDAI >= 10 or PUCAI > 10 with CRP > 0.5 mg/dl and/or FC >250 microg/g in a patient who previously responded to induction treatment.
Frequency of subtherapeutic IFX concentrations | 54 weeks
  Subtherapeutic IFX concentration is defined as IFX concentration at trough < 5 microg/ml (or <10 microg/ml in perianal CD) during maintenance treatment.
Frequency of Anti-Infliximab Antibodies | 54 weeks
  Evaluation of Anti-Infliximab Antibodies
Frequency of infusion reactions | 54 weeks
  Infusion reactions are defined as reactions that develop during the course of the infusion or within 1-2h of its completion.
Frequency of endoscopic remission | 54 weeks
  Endoscopic remission is defined in patients with Crohn's Disease as a Simple Endoscopic score for Crohn's Disease (SES-CD score) less than or equal to (<=) 2 and in patients with Ulcerative Colitis as a Mayo sub-score <= 1
Frequency of patients with treatment response at the end of induction between 12 and 14 weeks | Week 14
  Treatment response is defined as a decrease in PCDAI by 12.5 point or in PUCAI by 10 points with decrease in CRP by 50% compared to baseline
Frequency of patients with clinical remission at 14 weeks | Week 14
  Clinical remission is defined as PCDAI <10 or PUCAI <10
Frequency of clinical and biochemical remission at week 14 | Week 14
  Clinical and Biochemical remission is defined as PCDAI <10 or PUCAI <10 with CRP < 0.5 mg/dl and FC < 250 microg/g

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy